CLINICAL TRIAL: NCT03641911
Title: Incidence of Inadequate Pain Treatment in Ventilated Critically Ill Surgical Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Karuna Wongtangman, Instructor, Mahidol University
Other Study IDs: SI572/2017
Record Dates: First submitted 2017-11-08; First posted 2018-08-22 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Adult ICU Patients; Pain, Acute
Keywords: incidence; surgical ICU
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In SICU, Siriraj hospital there were no protocols place for the management of pain. All decisions were made according the attending physicians.

There were no information about incidence of inappropriate pain management in SICU due to lack of validated tool for assessment.

To date, Thai-version of BPS and CPOT were validated, the incidence of inappropriate pain management in SICU, Siriraj hospital should be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Expected duration of mechanical ventilation of more than 24 hours.

Exclusion Criteria:

* Quadriplegia.
* Receiving neuromuscular blocking medications.
* Coma or severe brain injury
* Neurosurgery/ CVT patients/ trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult surgical ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
overtreatment of pain (Richmond agitation sedation scale) | day0- 2 after admitted to ICU
  Richmond agitation sedation scale -3 to -5 undertreatment NRS 4-10 or CPOT 3-8
inadequate treatment of pain (Numeral rating scale) | day 0-2 after admitted to ICU
  Numeral rating scale 4-10 in communicable patient or critical care pain observation tool 3-8 in non-communicable patients

SECONDARY OUTCOMES:
Mortality rate | 30 days after admitted to ICU
ICU length of stay | 30 days after admitted to ICU
Duration of mechanical ventilation | 30 days after admitted to ICU
Incidence of acquired complication | 30 days after admitted to ICU
  * Ventilator associated pneumonia
  * GI hemorrhage
  * Venous thromboembolism
  * Central venous catheter colonization

CONTACTS AND LOCATIONS:
Locations (1):
- Karuna Wongtangman, Bangkok Noi, Bangkok, Thailand